CLINICAL TRIAL: NCT05628051
Title: Effect of Carotid Corrected Flow Time Combined With Perioperative Fluid Therapy on Preventing Hypotension After General Anesthesia Induction in Elderly Patients
Brief Title: Carotid Artery Corrected Flow Time as a Predictor of Hypotension After Induction of General Anesthesia in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022XHYG0018-01
Record Dates: First submitted 2022-11-17; First posted 2022-11-28 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: General Anesthesia Induction for Elective Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypotension after anesthetic induction group: Patients with hypotension after anesthetic induction
  Interventions: Procedure: ultrasonographic measurement of carotid artery corrected flow time (FTc)
- Non-hypotension after anesthetic induction group: Patients without hypotension after anesthetic induction
  Interventions: Procedure: ultrasonographic measurement of carotid artery corrected flow time (FTc)

INTERVENTIONS:
Procedure: ultrasonographic measurement of carotid artery corrected flow time (FTc) — Ultrasonic measurement of carotid corrected blood flow time: 1. Patient's head turned to the left 30°. Firstly, the 6.0 ~ 13.0MHz linear probe was placed longitudinally on the maternal neck, and the probe marker was oriented towards the maternal head. Real-time B-ultrasound images of the long axis of the right common carotid artery were obtained from the lower margin of the thyroid cartilage. Then, the probe was placed in the center of the carotid lumen, about 2cm from the bifurcation of the carotid artery, to obtain the arterial pulse Doppler flow spectrum and store the carotid flow waveform. 2. Using the caliper function of the ultrasonic instrument, carotid flow time (FT) was obtained by measuring the interval between the systolic ascending stage and the restroke notch. Wodey (W) formula to calculate FTc. FTc= FT+[1.29× (HR-60)

SUMMARY:
The number of elderly patients undergoing elective surgery has been growing in recent years. Elderly patients often have a variety of underlying diseases, including hypertension, coronary heart disease, diabetes, arteriosclerosis, etc., which increase the risk. When the elderly receive general anesthesia, hypotension often occurs after anesthesia induction. Once hypotension occurs, it may lead to myocardial ischemia, myocardial infarction, stroke and other serious complications. Therefore, in clinical anesthesia, a simple, quick and accurate prediction method is needed to evaluate and predict the risk of hypotension in elderly patients after induction, so that appropriate intervention measures can be taken in advance to reduce the incidence of hypotension in elderly patients after induction, thus reducing the occurrence of related complications and ensuring the safety of anesthesia and surgery.Carotid Artery Corrected Flow Time（FTc） is a recently developed volumetric predictor, which refers to the time between the the onset of systolic flow until the closure of the aortic valve. It is related to cardiac preload and can reflect cardiac output to a certain extent. It is considered as a reliable indicator for evaluating volume status and volumetric reactivity. Therefore, this study assessed the effect of FTc combined with perioperative fluid therapy on preventing hypotension after general anesthesia induction in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who received elective surgery under general anesthesia, aged 65-85 years old, gender unlimited, ASAI-II

Exclusion Criteria:

* uncontrolled hypertension
* unstable angina pectoris
* history of myocardial infarction
* after heart stent implantation
* severe arrhythmia：Atrial fibrillation、Ventricular premature beat, frequent atrial premature beat, other non-sinus rhythm
* pacemaker implants
* cardiomyopathy
* a left ventricular ejection fraction of < 40%
* history of neck trauma and surgery
* BMI>30

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who were scheduled to undergo elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Carotid artery corrected flow time (FTc) | 5 minutes before induction of general anesthesia
  the area under the receiver operating characteristics curve of corrected flow time in carotid artery measured by ultrasonography to predict hypotension after anesthetic induction

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Huang S, Liao Z, Chen A, Wang J, Xu X, Zhang L. Effect of carotid corrected flow time combined with perioperative fluid therapy on preventing hypotension after general anesthesia induction in elderly patients: a prospective cohort study. Int J Surg. 2024 Feb 1;110(2):799-809. doi: 10.1097/JS9.0000000000000863. PMID 37983823